CLINICAL TRIAL: NCT06754358
Title: Comparison of Perioperative Parameters of Femtosecond Laser-assisted Cataract Surgery Using Two Laser Systems: a Randomized Clinical Trial
Brief Title: Clinical Application Comparison of Two Femtosecond Laser Systems
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1312
Record Dates: First submitted 2024-12-15; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LenSx group (Active Comparator)
  Interventions: Procedure: LenSx
- Z8 group (Experimental)
  Interventions: Procedure: Z8

INTERVENTIONS:
Procedure: LenSx — Participants undergo FLACS using LenSx femtosecond laser system
  Arms: LenSx group
Procedure: Z8 — Participants undergo FLACS using Z8 femtosecond laser system
  Arms: Z8 group

SUMMARY:
The goal of this clinical trial is to compare the perioperative parameters of femtosecond laser-assisted cataract surgery (FLACS) using two laser systems.

Participants will:

Undergo FLACS using LenSx or Z8 femtosecond laser system Visit the clinic before the operation and 1 day, 1 week, and 1 month after the operation for checkups and tests Complete clinical measurements and dry eye questionnaires

ELIGIBILITY:
Inclusion Criteria:

1. Chinese Han patients aged 40 years or older
2. clinical diagnosis of age-related cataracts;
3. underwent FLACS with insertion of a posterior chamber IOL for the first eye.

Exclusion Criteria:

1. coexisting macular pathologies such as epiretinal membrane, macular hole or edema, or age-related macular degeneration. Patients with OCT scans of poor quality were excluded;
2. preoperative flare of more than 15ph/ms11, ECD<2000cells/mm2 or any other corneal pathologies;
3. coexisting serious ocular diseases including uveitis, uncontrolled glaucoma, optic atrophy , amblyopia, retinopathies, or inflammatory pathology of the eye;
4. history of intraocular trauma, surgery, or retinal laser procedures;
5. usage of systemic or topical steroids or NSAIDs within one month prior to surgery;
6. patients with diabetes or any other systemic diseases that might confound the results or increase the risk for postoperative inflammation;
7. intraoperative complications such as capsule tear, hyphema, vitreous loss, iris manipulation, or miosis after laser pre treatment requiring intracameral injection of epinephrine;
8. ocular conditions contraindicating FLACS including poorly dilated pupils (<5.0mm), narrow palpebral fissure, small hyperopic eyes with steep cornea (difficult to achieve suction), severe conjunctival chalasis, nystagmus, or lack of cooperation;
9. potentially pregnant women;
10. known sensitivity to concomitant medications used during perioperative period, participation in other clinical trial during the time of visit, or poor cooperation in diagnostic tests or non-compliance at follow-up.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
ocular staining score | 1 month after operation
  The ocular staining score ranged from 0 to 12. A score of 0 indicated no corneal or conjunctival staining with fluorescein or lissamine green dye, respectively. A score of 12 indicated severe staining of the cornea and conjunctiva with confluent and central fluorescein staining, the presence of corneal filaments, and confluent areas of lissamine green of the bulbar conjunctiva of greater than or equal to 4 mm2.

SECONDARY OUTCOMES:
ocular staining score | 1 day and 1 week after operation
  The ocular staining score ranged from 0 to 12. A score of 0 indicated no corneal or conjunctival staining with fluorescein or lissamine green dye, respectively. A score of 12 indicated severe staining of the cornea and conjunctiva with confluent and central fluorescein staining, the presence of corneal filaments, and confluent areas of lissamine green of the bulbar conjunctiva of greater than or equal to 4 mm2.
phacoemulsification time | in the operation
ultrasound power | in the operation
vacuum docking time | in the operation
femtosecond laser emission time | in the operation
femtosecond laser-assisted capsulorhexis time | in the operation
femtosecond laser-assisted pre-chop time | in the operation
surgical time | in the operation
surgical complication | in the operation
DEQ-5 questionnaire | 1 week and 1 month after the operation
  The dry-eye questionnaire-5 (DEQ-5) is a validated questionnaire that has been shown to discriminate between different severities of dry eye. Participants self-assessed the frequency and severity of eye discomfort, eye dryness, and watery eyes experienced during the evening of a typical day within the last month. Responses were given using a Likert scale with scoring criteria from 0 = never experienced the symptom to 5 = extremely severe experience of symptom. The sum of the scores from the five questions was used in the analysis.
OSDI questionnaire | 1 week and 1 month after the operation
  Ocular surface disease index (OSDI) is a widely accepted questionnaire on subjective symptoms in patients with dry eyes. It consisted of 12 questions on eye-related symptoms, vision-related function, and environment-related symptoms. Each question is evaluated according to the frequency of occurrence: never, 0 point; occasionally, 1 point; often, 2 points; most of the time, 3 points; all the time, 4 points. Not all the 12 questions needed to be answered. If the question is that the patient didn't participate in the activity or the environment that would not be in the case, it would not be answered and scored. The final score is calculated according to the formula: OSDI values=(sum of all survey items)×100/(answered survey items)×4.
tear meniscus height | 1 day, 1 week, and 1 month after the operation
  The tear meniscus assessment height was measured with the Ocular Surface Analyser (SBM Sistemi, Orbassano, Italy)
noninvasive tear film breakup time | 1 day, 1 week, and 1 month after the operation
  Noninvasive tear film breakup time was assessed automatically using the Ocular Surface Analyser (SBM Sistemi, Orbassano, Italy). The participants were instructed to blink naturally two times and then to cease blinking until instructed to blink again. Three measurements were performed for each eye and the average for each eye included for analysis.
tear-film assessment | 1 day, 1 week, and 1 month after the operation
  The tear-film assessment was assessed with the Ocular Surface Analyser (SBM Sistemi, Orbassano, Italy).
Schirmer I test | 1 day, 1 week, and 1 month after the operation
  The Schirmer I test was carried out under natural light. A 5 mm×35 mm Schirmer test strip was placed in the middle and outer 1/3 junction of the lower conjunctival sac of the affected eye without anesthesia. The patient was asked to close eyes gently. After 5min, the strip was removed and the wet length of the strip was measured. Values less than 5 mm are indicators for dry eye syndrome.
visual acuity | 1 day, 1 week, and 1 month after the operation
intraocular pressure | 1 day, 1 week, and 1 month after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China